CLINICAL TRIAL: NCT05942443
Title: Treatment of Trigger Finger With Metacarpophalangeal Joint Blocking Orthosis Versus Relative Motion Extension Orthosis
Brief Title: Comparative Effectiveness of the Two Splints in Trigger Finger
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Cigdem Ayhan, professor doctor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-772.02-2507
Record Dates: First submitted 2023-06-13; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Trigger Finger
Keywords: Trigger finger; relative motion splint; pain; function; satisfaction; static splint
MeSH Terms: conditions — Trigger Finger Disorder; Pain; Personal Satisfaction | interventions — Treatment Expectations; Aftercare

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned in a 1:1 ratio to either the MCP-blocking orthosis group or the RME orthosis group, using a simple random sampling method.
Masking Description: Splints are fabricated by the orthotist and outcome assessments are performed by a physiotherapist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCP blocking orthosis (Active Comparator): Patients received the MCP blocking orthosis
  Interventions: Procedure: Pre-treatment; Procedure: Post-treatment
- RME orthosis (Experimental): Patients received the RME orthosis for six weeks
  Interventions: Procedure: Pre-treatment; Procedure: Post-treatment

INTERVENTIONS:
Procedure: Pre-treatment — The custom MCP blocking orthosis was made of a 1.6-mm-thick thermoplastic material that extends from the palm over the MCP joint and includes a ring around the proximal phalanx. It is designed to block the MCP joint in flexion of 10°-20° while allowing full range of motion of the proximal and distal interphalangeal joints.
Procedure: Post-treatment — The RME orthosis was fabricated from 3.2-mm-thick thermoplastic material with the affected finger positioned at an extension of approximately 10°-20° relative to the adjacent fingers.

SUMMARY:
RME orthosis is recommended for the treatment of trigger finger. However, its efficacy has not been studied in trigger finger patients. Given the increasing popularity of this orthosis among clinicians, it is important to evaluate their effectiveness to provide evidence for its use in trigger finger. The purpose of this study was to compare the efficacy of a 6-week orthotic intervention in a randomly selected group of patients with trigger finger using MCP-blocking and RME orthoses.

DETAILED DESCRIPTION:
Generally, three types of orthoses are used in the treatment of trigger finger. Some authors used MCP blocking orthosis, while others used DIP or PIP blocking orthosis. Comparative studies are quite limited, as only one study comparing two orthotic designs found that the MCP blocking orthosis was more effective than the DIP blocking orthosis.The MCP blocking orthosis, which restricts the MCP joint to 10-15° of flexion, is commonly used in the conservative treatment of trigger finger.An RME orthosis could be an alternative orthotic treatment option for trigger finger because it holds the MCP in an extended position. The RME orthosis is thought to prevent flexion of the affected finger, thereby limiting tendon glide. This reduces the pressure on the A1 pulley, allowing the tendon to glide more smoothly, reducing the likelihood of triggering. Despite limiting motion,the orthosis still allows the patient to perform daily activities with the orthosis. Therefore, positioning the MCP joint in extension could provide additional benefits in trigger finger. The relative motion orthosis is a new orthotic design that positions the affected finger in 10-15 degrees of extension relative to the adjacent fingers.It also has several advantages, including small size, low-profile design, easy and inexpensive fabrication, and better patient compliance. The primary objective of this study was to compare the efficacy of a 6-week orthotic intervention for pain relief in a randomly selected group of patients with TF using the MCP blocking orthosis and the RME orthosis. The secondary objective was to determine the comparative effectiveness of the orthoses on function and satisfaction with the orthosis.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with Stage 1-3 trigger finger (Froimson Classification)
* A1 pulley triggering

Exclusion Criteria:

* trigger thumb
* multiple trigger fingers on one hand
* neurological disorders
* rheumatologic diseases
* pregnancy
* patients who had received a steroid injection in the affected finger within the previous six months
* patients who had previously undergone trigger release surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Finger Pain | baseline, sixth week
  Numeric Pain Rating Scale (NPRS)

SECONDARY OUTCOMES:
Satisfaction with the orthosis | sixth week
  The Quebec Assistive Technology User Satisfaction Evaluation (Quest 2.0)
Hand Function | baseline, sixth week
  Disabilities of Arm, Shoulder, and Hand Questionnaire (DASH)

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Faculty of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT05942443/Prot_SAP_000.pdf